CLINICAL TRIAL: NCT03943810
Title: Characterizing ER Activities for Failure Prevention
Brief Title: Analysis and Improvising Working Practices in the ER
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Dr. Yahel Giat (Unknown); Pr. Merav Lidar (Unknown); Dr. Michael Dreyfuss (Unknown); Dr. Avinoah Irony (Unknown); Dr. Gabrieal Breuer (Unknown)
Responsible Party: Principal Investigator, Dr. Eitan Giat, Principal investigator, senior reumatologist in the rheumatology unit, Sheba Medical Center
Other Study IDs: 5132-18-SMC
Record Dates: First submitted 2019-05-05; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: EMERGENCY MEDICINE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
Analysis of electronic files of patients presenting to the emergency department to improve current practice

DETAILED DESCRIPTION:
Overcrowding in the emergency department (ED) is a pressing healthcare issue globally and has been shown to negatively affect the quality of treatment, clinical outcomes and patient satisfaction.

In recent years, an increasing number of studies have tried to implement changes in the ED to increase efficiency and thereby reduce the length of stay (LOS). Examples to these efforts include physician triage, expanding the nursing scope of practice and patient-flow design (e.g., creating fast track units) in the ED. Importantly, not all intuitive changes in the ED resulted in the reduction of LOS Therefore, implementing changes in the ED must be done with caution and preceded with a cost-benefit analysis of the effects of the intervention using available retrospective data.

This research was conducted in the ED of Sheba Medical Center (SMC), a tertiary government-owned hospital in Israel with 1400 beds. This study is a retrospective medical record review of patients admitted to the adult primary SMC ED. The study sample comprises all the walk-in patients that visited the ED between January 2013 and December 2017. The data here does not include other EDs located elsewhere in SMC, (e.g., pediatric ED, gynecology ED, ophthalmology ED, and psychiatric ED). All admissions files in SMC ED are recorded in a computerized system with negligible exceptions (such as power outage and connection or server maintenance). The time and date of every change in the electronic files are also recorded in the system. Therefore, it is possible to track the waiting times as well as the full content of the admission file.

The aim of this study is to identify and analyze potential modifications in current ED practice which may improve outcomes such as LOS, missed diagnosis, leaving without being seen, patient satisfaction, etc.

ELIGIBILITY:
Inclusion Criteria:

* all the patients that visited the SMC - ED between August 2014 and December 2017

Exclusion Criteria:

* patients in which the electronic file is absent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the patients admitted to the adult primary SMC ED ED between August 2014 and December 2017.
  . The data here did not include other EDs located elsewhere in SMC, (e.g., pediatric ED, gynecology ED, ophthalmology ED and psychiatric ED).
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | Starting from January1st 2014 until January 30th 2018
  The time between admitting the patient to the ED and the time of decision to release or admit to hospital
left without being seen | Starting from January1st 2014 until January 30th 2018
  amount of patients who leave the ED without being seen by a physician
missed diagnosis | Starting from January1st 2014 until January 30th 2018
  Change of preliminary diagnosis made by ED physician compared to diagnosis after admission to hospital, or after readmission to ED
physician mistakes | Starting from January1st 2014 until January 30th 2018
  Errors made by ED physician in the management of patients in the ED
Admission to hospital | Starting from January1st 2014 until January 30th 2018
  The rate of hospitalization compred to the rate of discharge from ED
return to ED after discharge | Starting from January1st 2014 until January 30th 2018
  patients returning to hospital within 30 days of discharge from ED
Time till being seen by a physician | Starting from January1st 2014 until January 30th 2018
  We measure the time it took for the patient to be seen by an ED physician

IPD SHARING:
Plan to Share IPD: No
all data is encrypted and unidentified